CLINICAL TRIAL: NCT02251561
Title: Clinical Evaluation of Opti-Free III Compared to Opti-Free Plus®
Brief Title: Clinical Evaluation of Opti-Free III (FID 109182) Compared to Opti-Free Plus® in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: CVKK2013-01
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Corneal Staining
Keywords: contact lenses; contact lens solution; corneal staining; fluorescein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 109182 (Experimental): Senofilcon A contact lens pre-soaked in FID 109182 worn in the right or left eye as randomized for 2 hours
  Interventions: Device: FID 109182; Device: Senofilcon A contact lens
- Opti-Free Plus (Active Comparator): Senofilcon A contact lens pre-soaked in Opti-Free Plus worn in the fellow eye for 2 hours
  Interventions: Device: Opti-Free Plus; Device: Senofilcon A contact lens

INTERVENTIONS:
Device: FID 109182 — Investigational multipurpose contact lens cleaning and disinfecting solution
  Other Names: Opti-Free III
  Arms: FID 109182
Device: Opti-Free Plus — Commercially available multipurpose contact lens cleaning and disinfecting solution
  Other Names: Opti-Free Plus®
  Arms: Opti-Free Plus
Device: Senofilcon A contact lens — Commercially available silicone hydrogel contact lens
  Other Names: Acuvue® Oasys®

SUMMARY:
The purpose of this study is to compare an investigational contact lens care product (FID 109182) to a commercially available contact lens product (Opti-Free Plus®) for corneal staining when used with Acuvue® Oasys® contact lenses. The contact lenses will be pre-soaked in the products for 24-48 hours prior to a 2-hour contralateral wear period.

ELIGIBILITY:
Inclusion Criteria:

* Soft contact lenses habitual wearer, both eyes.
* Voluntarily sign Informed Consent.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Unable to tolerate the ingredients in Opti-Free® and similar contact lens care products.
* Potential use of eye drops during the study, including over-the-counter products, except for artificial tear eye drops.
* Eye infection, blepharitis, iris inflammation, or severe eye inflammation.
* Corneal staining greater than Grade 1 at baseline.
* Pregnant, lactating, or intend to become pregnant during study period.
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsunemitsu Senta, Study Director — Alcon Japan, Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from one study site located in Japan.
Pre-assignment Details: Of the 36 subjects enrolled in the study, 8 were exited prior to product exposure [did not meet eligibility criteria (5), and subject withdrawal (3)]. This reporting group includes all subjects who used the study products (28).
Groups:
- FID 109182/Opti-Free Plus: Senofilcon A contact lens pre-soaked in FID 109182 in 1 eye, with senofilcon A contact lens pre-soaked in Opti-Free Plus in the fellow eye. Lenses worn contralaterally for 2 hours.
Period: Overall Study
Arm/Group | FID 109182/Opti-Free Plus
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who used the study products.
Arm/Group | FID 109182/Opti-Free Plus
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Region of Enrollment [Number; unit: participants]
  Japan | 28

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Scoring ≥ 2 for Corneal Staining Density With Fluorescein
Description: The contact lens was removed, the cornea was stained with fluorescein (ophthalmic dye), and pictures of the corneal surface were taken. Corneal staining density was evaluated for each eye individually against representative pictures and scored on a 0-3 scale (0=No staining; 1=Staining with low density; 2=Staining with moderate density; 3=Staining with severe density). Proportion of participants is reported as a percentage.
Time Frame: Day 1, after 2 hours of wear
Population: This analysis population includes all subjects who used the study products and had examination/observation data after use.
Measure: Number; unit: percentage of participants
Groups:
- FID 109182: Senofilcon A contact lens pre-soaked in FID 109182 worn in 1 eye for 2 hours
- Opti-Free Plus: Senofilcon A contact lens pre-soaked in Opti-Free Plus worn in 1 eye for 2 hours
Arm/Group | FID 109182 | Opti-Free Plus
Number analyzed (Participants) | 27 | 27
percentage of participants | 92.6 | 22.2

2. Secondary Outcome: Proportion of Participants Scoring ≥ 2 for Corneal Staining Area With Fluorescein
Description: The contact lens was removed, the cornea was stained with fluorescein (ophthalmic dye), and pictures of the corneal surface were taken. Corneal staining area was evaluated for each eye individually against representative pictures and scored on a 0-3 scale [0=No staining; 1=Staining with small area (1 to 25% of corneal surface); 2=Staining with medium area (26 to 50% of corneal surface); 3=Staining with large area (51% of corneal surface or greater)]. Proportion of participants is reported as a percentage.
Time Frame: Day 1, after 2 hours of wear
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FID 109182 | Opti-Free Plus
Number analyzed (Participants) | 27 | 27
percentage of participants | 92.6 | 44.4

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: This analysis population includes all subjects who used the study products. In this contralateral study, number at risk is presented by eye.
Arm/Group | FID 109182 | Opti-Free Plus
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.